# **ABBOTT**

# **Statistical Analysis Plan**

# Module 1 (Non-standard data and analyses)

Version 2.0, Date 06 Aug 18

Study: RACE3003

Multicenter, open-label, controlled, randomized clinical study to evaluate the efficacy and safety of Racecadotril in infants, children and adolescents with acute diarrhea





# TABLE OF CONTENTS

| SIGNA | TURE PAGE | 2 |
|------------|-----------------------------------------------------------|----|
| 1. | ABBREVIATIONS | 5 |
| 1.1 | Standard Abbreviations | 5 |
| 2. | Introduction | 7 |
| 3. | SUMMARY OF THE PROTOCOL | 8 |
| 3.1 | Overall Study Plan | |
| 3.2 | Study Flowchart | |
| 3.3 | Study Objectives | |
| 4. | STATISTICAL ANALYSIS | 12 |
| 4.1 | Subject samples | 12 |
| 4.2 | Efficacy analysis | 12 |
| 4.2.1 | Primary Efficacy Analysis | 12 |
| 4.2.2 | Secondary efficacy analysis | 14 |
| 4.2.3 | Other efficacy analysis | 16 |
| 4.3 | Safety analysis | 16 |
| 4.4 | Interim Analysis | 18 |
| 4.5 | Data Safety Monitoring Board | 18 |
| 4.6 | Safety Management Team | 19 |
| 5. | DESCRIPTION OF NON-STANDARD DATA COLLECTED AND | |
| | DERIVED VARIABLES | |
| 5.1 | Other Non-Standard Baseline Characteristics | |
| 5.2 | Non-Standard Disease History | |
| 5.3 | Efficacy data | |
| 5.4 | Non-standard Safety Data | |
| 5.5 | Drug Accountability and Exposure | |
| 5.5.1 | Drug Accountability | |
| 5.5.2 | Exposure | 22 |
| 6. | FURTHER SPECIFICATIONS TO THE STANDARD ANALYSES | |
| <i>c</i> 4 | MODULE 2 | |
| 6.1 | Trial Design [2] | |
| 6.1.1 | Trial Periods | |
| 6.1.2 | Trial Elements | |
| 6.1.3 | Trial Arms | |
| 6.1.4 | Visits and related definitions | |
| 6.2 | Further Specifications to the Standard Tables in Module 2 | |
| 6.3 | Other Further Specifications | 26 |

| 7. | CHANGES TO PLANNED ANALYSES | 27 |
|-----|-----------------------------|----|
| 8. | REFERENCE | 28 |
| 9. | APPENDICES | 29 |
| 9.1 | Study Flowchart | |

#### 1. ABBREVIATIONS

#### 1.1 Standard Abbreviations

AE adverse event

ANCOVA analysis of covariance

ATC Anatomical Therapeutic Chemical (class)

AUC area under the curve
BDR blind data review
bpm beats per minute
CRF case report form

CRO contract research organization

CV coefficient of variation
DBP diastolic blood pressure
DDT data definition table

DSMB data safety monitoring board

ECG electrocardiogram FA Full Analysis

FDA food and drug administration

Geo. mean geometric mean

GOP global standard operating procedure

HLGT High Level Group Term

HLT High Level Term

ICH International Conference on Harmonization
LDA day number of the last day of drug administration

LLOQ lower level of quantification

LLT Lowest Level Term

LOCF last observation carried forward

max maximum

MedDRA Medical Dictionary for Regulatory Activities

min minimum

N,n number of observations

NA not applicable
OC observed cases
PD pharmacodynamic
PK pharmacokinetic
PP Per Protocol
PT Preferred Term
QOL quality of life

SAE serious adverse event
SAP statistical analysis plan
SBP systolic blood pressure
SD standard deviation
S.I. System International
SOC System Organ Class

SOP standard operating procedure

TARC Therapeutic Area Review Committee
TEAE treatment-emergent adverse event

TESAE treatment-emergent serious adverse event

TLF/T,L,F tables, listings and figures
ULOQ upper limit of quantification
URL upper reference limit

URL upper reference limit WC windowing convention

WHO-DD(E) World Health Organization – Drug Dictionary (enhanced)

# 2. Introduction



#### 3. SUMMARY OF THE PROTOCOL

#### 3.1 Overall Study Plan

This is a controlled, open-label, parallel-group study evaluating the efficacy and safety of Racecadotril in infants, children and adolescents with acute diarrhea. The number of subjects to be screened is 150 in order to enroll 124 subjects for either standard treatment (oral rehydration solution, ORS) alone or ORS plus Racecadotril.

1.5 mg/kg of Racecadotril will be administered, 3 times daily, via the oral route. Study drug intake will start either with the noon or the evening dose on day 1.

In infants less than 9 kg: one 10 mg sachet 3 times daily.

In infants from 9 kg to <13 kg: two 10 mg sachets 3 times daily.

In children from 13 kg to 27 kg: one 30 mg sachet 3 times daily.

In children from more than 27 kg to 60 kg: two 30 mg sachets 3 times daily.

In children or adolescents of 60 kg or higher: 100 mg capsule 3 times daily

Standard treatment is oral rehydration solution (ORS) according to the registered local label and the instruction of the investigator. The same brand of ORS and the same age-appropriate standardized treatment pattern for the subjects will be applied throughout the trial. ORS treatment and dosing will be documented in the CRF.

#### **Screening and Enrolment (Day 1, Visit 1)**

Subjects presenting with acute diarrhea will be evaluated for eligibility. They will undergo a physical examination including assessment of dehydration level, vital signs, a review of their medical history and concomitant medication. If the subjects are eligible for the study, demographics, number of stools during the last 24 hours will be assessed as baseline values. The subjects will be randomized to Racecadotril plus ORS or ORS alone. On Day 1 the subject will start with study treatment. The starting dose will either be the noon or the evening dose depending on the timing of Visit 1.

#### Treatment period (until recovery, maximally 5 days)

Subjects will be treated with Racecadotril tid according to the body weight dose requirement on an in- or out-patient basis for maximum 5 days. One arm will be treated with ORS alone as standard treatment, the other treatment arm will be treated with ORS (according to the registered local label and the instruction of the investigator) in addition to Racecadotril. ORS will be prescribed by the investigator and will be taken according to the product label and the instruction of the investigator. The parent(s)/caregiver(s) will be instructed to stop study drug treatment when the patient recovered. On each day, the parent(s)/caregiver(s) will fill in their diaries, documenting the date and time of each individual stool, the stool consistency of each stool (diarrheal/watery or normal), the amount of ORS and the study drug intake. After the occurrence of two consecutive normal stools, the parent(s)/caregiver(s) can stop recording of the diary and return to the study site for the end of treatment visit. The date of recovery is the day when the first of two consecutive normal stools were excreted. AEs are to be reported on an ongoing basis.

# End of treatment (Day 6 or early recovery, Visit 2)

The last dose of study drug will be the morning dose of day 6, if not recovered earlier. The same day, or within 24 hours after recovery, the parent(s)/caregiver(s) will visit the site for the end of treatment visit of the child. Data on vital signs, AEs, physical examination and concomitant medication will be collected. Subjects will return their diaries and unused medication.

#### Safety follow-up

A phone call will be performed at 5-7 days after end of the treatment period for the safety follow-up.



Figure 3-1 Study design

#### 3.2 Study Flowchart

The flowchart of the study can be found in Appendix 9.1.

#### 3.3 Study Objectives

#### **Primary Objective(s)**

The primary objective is to evaluate the efficacy of Racecadotril in addition to standard treatment oral rehydration solution (ORS) versus ORS alone in infants, children and adolescents (3 months until <18 years) with acute diarrhea measured as duration of diarrhea (hours) between the start of treatment until final diarrheal/watery stool before recovery or end of study treatment (treatment duration maximal 5 days).

Duration of diarrhea is defined by date and time of the evacuation of the final watery/diarrheal stool before recovery derived from the daily diary (see Figure 3-2 Duration of diarrhea and Time until recovery definition).



Figure 3-2 Duration of diarrhea and Time until recovery definition

#### Secondary Objective(s)

- Number of recovered subjects per treatment group in total and until each individual treatment day. Mean and median time until recovery per treatment group.
- Time until recovery, defined by date and time of the evacuation of the first of two consecutive normal stools or no stool within 12 hours after first normal stool (see Figure 3-2 Duration of diarrhea and Time until recovery definition).
- Global Physician Assessment at the end of treatment:
  - o 1 = Complete relief of acute diarrhea,
  - $\circ$  2 = marked improvement of acute diarrhea,

- o 3 = moderate improvement of acute diarrhea,
- o 4 = slight improvement of acute diarrhea,
- $\circ$  5 = no change in acute diarrhea,
- o 6 =worsening of acute diarrhea. (Treatment success = GPA score of 1 or 2).
- For toilet trained children and adolescents: number of stools per day as well as number of watery stools per day from start of treatment and until end of study treatment.

#### Safety Objective(s)

To evaluate the safety and tolerability of Racecadotril together with oral rehydration solution (ORS) versus ORS alone in infants, children and adolescents with acute diarrhea by adverse events, physical examination and vital signs.

#### 4. STATISTICAL ANALYSIS

#### 4.1 Subject samples

There will be five subject samples.

- The all subjects consented sample will consist of all subjects who:
  - Gave their informed consent.
- The all subjects allocated to treatment sample will consist of all subjects who:
  - Were in the all subjects consented sample; and
  - Were allocated to treatment.
- The safety sample will consist of all subjects who:
  - Were in the all subjects allocated to treatment sample; and
  - Had at least one dose of study medication administered.
- The full analysis (FA) sample will consist of all subjects who:
  - Were included in the safety sample; and
  - Had data for at least one post-baseline assessment of any efficacy measurement.
- The per-protocol (PP) sample will be defined through blind data review and will consist of all subjects who:
  - Were included in the FA sample; and
  - Did not present any major protocol violation (consideration about exclusion of patients from *the PP sample* will be performed at the Blind Data Review).

#### 4.2 Efficacy analysis

The *FA subject sample* will be used for the analysis of the efficacy data. Additionally, primary efficacy results analysis will be conducted on the *PP sample* as the sensitivity analysis. Descriptive statistics will be presented by treatment arm and by stratification level (Age Category) for all planned efficacy endpoints.

All analyses will be based on available data only and no missing data will be imputed.

All parameters will be summarized using descriptive statistics and listed.

#### 4.2.1 Primary Efficacy Analysis

The primary efficacy variable is the duration (hours) of diarrhea (treatment duration max 5 days). Duration of diarrhea is defined by date ("event" date) of the evacuation of the last diarrheal/watery stool before recovery.

In order to compare the primary efficacy parameter, duration of diarrhea, between the treatment groups, a Kaplan Meier (KM) analysis will be performed. The KM algorithm will be applied to derive the median duration and the 95% confidence intervals for the median, Q1, Q3 and mean duration with Greenwood's estimator of standard deviation of Kaplan-Meier estimator.

The log-rank test will be used to test whether the difference between the duration of diarrhea between two treatment groups is statistically significant, i.e. p-value <0.05.

For duration estimation the date and time of first drug intake will be assumed as start time point and all subjects without "event" will be censored by 6 days (144 hours).

```
SAS code for the analysis:
```

```
PROC LIFETEST DATA = [dataset name]

METHOD=KM PLOTS=SURVIVAL

OUTSURV=SURV CONFTYPE=LOGLOG ATRISK;

TIME [time variable]*[censor variable];

STRATA [arm variable];

RUN;
```

The "OUTSURV" statement provides variables that contains the lower and upper limits of the pointwise confidence intervals for the survivor function ("SDF\_LCL" and "SDF\_UCL"), this confidence intervals should be transformed for tables as follows:

```
[Lower limit var name] = round(100*(1-SDF_UCL),.1);
[Upper limit var name] = round(100*(1-SDF_LCL),.1);
```

As a first sensitivity analysis, duration of diarrhea will be analyzed by age subgroups as follows:

- Racecadotril + ORS (age subgroup 3 to < 24 month) vs ORS (age subgroup 3 to < 24 month) comparison;
- Racecadotril + ORS (age subgroup >= 2 to <12 years) vs ORS (age subgroup >= 2 to <12 years) comparison;
- Racecadotril + ORS (age subgroup 12 to < 18 years) vs ORS (age subgroup 12 to < 18 years) comparison;

As a second sensitivity analysis, duration of diarrhea will be analyzed by weight/dosing subgroups as follows:

• Racecadotril + ORS (Infants less than 9 kg) vs ORS (Infants less than 9 kg) comparison;

- Racecadotril + ORS (Infants from 9 kg to < 13 kg) vs ORS (Infants from 9 kg to < 13 kg Infants from 9 kg to < 13 kg) comparison;
- Racecadotril + ORS (Children from 13 kg to 27 kg) vs ORS (Children from 13 kg to 27 kg) comparison;
- Racecadotril + ORS (Children from more than 27 kg to 60 kg) vs ORS (Children from more than 27 kg to 60 kg) comparison;
- Racecadotril + ORS (Children or adolescents of 60 kg or higher) vs ORS (Children or adolescents of 60 kg or higher) comparison;

```
SAS code for the analysis:
```

```
PROC LIFETEST DATA = [dataset name]

METHOD=KM PLOTS=SURVIVAL

OUTSURV=SURV CONFTYPE=LOGLOG ATRISK;

TIME [time variable]*[censor variable];

STRATA [arm variable];

BY [age subgroup variable];

RUN;
```

PROC LIFETEST DATA = [dataset name]

METHOD=KM PLOTS=SURVIVAL

OUTSURV=SURV CONFTYPE=LOGLOG ATRISK;

TIME [time variable]\*[censor variable];

STRATA [arm variable];

BY [weight/dosing category variable];

RUN;

Description of the Cox regression model analysis is presented in the Section 4.2.3 of the SAP.

#### 4.2.2 Secondary efficacy analysis

The secondary efficacy variables are

- Number of recovered subjects per treatment group in total and until each individual treatment day. Mean and median time until recovery per treatment group.
- Time until recovery, defined by date and time of the evacuation of the first of two consecutive normal stools.

Time until recovery, number of recovered subjects per treatment group in total and until each individual treatment day and mean and median time until recovery per treatment group will be estimated Kaplan Meier analysis as described for the primary endpoint.

- Global Physician Assessment at the end of treatment:
  - o 1 = Complete relief of acute diarrhea,
  - $\circ$  2 = marked improvement of acute diarrhea,
  - o 3 = moderate improvement of acute diarrhea,
  - o 4 = slight improvement of acute diarrhea,
  - $\circ$  5 = no change in acute diarrhea,
  - o 6 =worsening of acute diarrhea.

Frequencies table will be performed for the Global Physician Assessment at the end of treatment by GPA score and by success rating. Treatment will be rated as success when the GPA score equals 1 or 2.

Description of the subgroup analysis is presented in the Section 4.2.3 of the SAP.

The comparisons of treatment arms using Fisher exact test will be performed by proportion of patients with Global Physician Assessment success at the end of treatment.

SAS code for the analysis:

```
PROC FREQ DATA = [dataset name];
WEIGHT [GPA frequency] / ZEROS;
TABLES [GPA yes/no level] * [Arm] / EXACT FISHER;
RUN;
```

If SAS code produces the "Row or column sum zero. No statistics computed for this table." output due to insufficient memory available to complete the Fisher exact computations, then the p-value should be assumed as equal 1.0000.

• For toilet trained children and adolescents: number of stools per day as well as number of watery stools per day from start of treatment and until end of study treatment.

Number of stools and number of watery stools will be presented descriptively per treatment group and cumulatively until each day of treatment.

#### 4.2.3 Other efficacy analysis

Additionally, duration of diarrhea and time to recovery will be analyzed using Cox regression model where treatment group, age group, and dosing/weight group will be included as covariates. Relative risk will be presented for each covariate with 95% confidence intervals (Relative risk is referred to as "Hazard ratio" in the output from PROC PHREG SAS procedure).

SAS code for the analysis:

```
PROC PHREG DATA = [dataset name];

CLASS [arm variable] (ref=[reference level])

[age group] (ref=[reference level])

[weight/dosing category] (ref=[reference level]);

MODEL [time variable] * [censor variable] =

[arm variable] [age group] [weight/dosing category] / RL;
```

RUN;

The results of the exploratory analyses using Cox regression model will be provided in appropriate tables with the main results (see 10.1.4.1.2.1; 10.1.4.1.2.2; 10.1.4.1.5.1; 10.1.4.1.5.2; 10.1.4.2.2.1 and 10.1.4.2.2.2 table shells).

The comparisons by subgroup for GPA score success rating using Fisher exact test will be performed using the following SAS code:

```
PROC FREQ DATA = [dataset name];
WEIGHT [GPA frequency] / ZEROS;
TABLES [GPA yes/no level] * [Arm] / EXACT FISHER;
BY [age subgroup variable];
RUN;
```

If SAS code produces the "Row or column sum zero. No statistics computed for this table." output due to insufficient memory available to complete the Fisher exact computations, then the p-value should be assumed as equal 1.0000.

The results of the exploratory analyses will be provided in appropriate tables with the main results (see Table 10.1.4.2.3), no adjustment for multiplicity will be done due to the exploratory nature of analyses.

#### 4.3 Safety analysis

The Safety Sample will be used for the analysis of the safety and tolerability data.

Descriptive statistics for all safety and tolerability data will be presented by treatment arm and by stratification level (Age Category).

AEs are considered treatment emergent (TE) if they start or worsen at or after the first administration of study drug and before or on the day of last administration of study drug plus a gap period of 1 day (24 hours).

AEs will be reported on a per-subject basis, i.e. counting subjects rather than events. This means that if a subject suffers the same AEs repeatedly during the applicable study period, the event will be counted only once for that period. Repeated events per subject will be summarized according to the following rule: if a subject suffered the same AE more than once, the event will be assigned the worst severity, the closest relationship to the study drug and the earliest starting date. Only treatment emergent AEs will be reported. In the listings, however, all occurrences of the AEs will be presented.

For each unique treatment, treatment emergent AEs will be summarized per primary SOC, per HLT by primary SOC and per PT by HLT and primary SOC. Severity and drug-event relationship of treatment emergent AEs are summarized separately. Non-TEAEs will be listed.

Vitals signs: Height (m), Weight (kg), Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Pulse (bpm), including changes from baseline will be summarized. A frequency table will be presented for markedly abnormal values (presented in the table categories includes "to high", "to low" and "normal" levels based on normal ranges).

Temperature data will be presented in appropriate listing only.

RACE3003 clinical study was conducted with the involvement of local laboratories, thus local normal ranges have been used in each particular site (the ranges are presented below). Additional footnote ("Created *<table/listing>* based on site specific ranges.") will be presented for appropriate tables and listings in the statistical analysis report.

| | Normal Heart Rate by Age (beats/minute) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Age | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| 1-12 month | 100-140 | 100-190 | 100-190 | 100-160 | 100-190 | 100-190 | 110-170 | 100-190 | 100-190 |
| 1-3 years | 98-120 | 98-140 | 95-110 | 98-140 | 98-140 | 98-140 | 100-130 | 98-140 | 98-140 |
| 3-6 years | 80-105 | 80-120 | 80-120 | 80-120 | 80-120 | 80-120 | 85-115 | 80-120 | 80-120 |
| 6-9 years | 75-90 | 75-118 | 75-110 | 75-118 | 75-118 | 75-118 | 75-105 | 75-118 | 75-118 |
| 9-12 years | 70-90 | 60-100 | 60-100 | 60-100 | 60-100 | 60-100 | 70-90 | 60-100 | 60-100 |
| 12-18 years | 70-90 | 60-100 | 60-100 | 60-100 | 60-100 | 60-100 | 70-90 | 60-100 | 60-100 |

| | Normal Systolic Blood Pressure by Age (mm Hg) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Age | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| 1-12 month | 80-112 | 90-112 | 85-105 | 90-112 | 90-112 | 90-112 | 75-80 | 90-112 | 90-112 |
| 1-3 years | 90-112 | 100-112 | 85-110 | 100-112 | 100-112 | 100-112 | 80-85 | 100-112 | 100-112 |
| 3-6 years | 100-116 | 100-116 | 85-115 | 100-116 | 100-116 | 100-116 | 90-95 | 100-116 | 100-116 |
| 6-9 years | 100-122 | 100-122 | 95-120 | 100-122 | 100-122 | 100-122 | 95-105 | 100-122 | 100-122 |
| 9-12 years | 100-126 | 110-126 | 110-125 | 110-126 | 110-126 | 110-126 | 105-115 | 110-126 | 110-126 |

| | Normal Systolic Blood Pressure by Age (mm Hg) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Age | | | | | | | | | |
| 12-18 years | 110-120 | 110-136 | 110-130 | 110-136 | 110-136 | 110-136 | 110-120 | 110-136 | 110-136 |

| | Normal Diastolic Blood Pressure by Age (mm Hg) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Age | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| 1-12 month | 50-74 | 50-74 | 45-60 | 50-74 | 50-74 | 50-74 | 50-74 | 50-74 | 50-74 |
| 1-3 years | 60-74 | 60-74 | 50-60 | 60-74 | 60-74 | 60-74 | 50-55 | 60-74 | 60-74 |
| 3-6 years | 60-76 | 60-76 | 55-60 | 60-76 | 60-76 | 60-76 | 50-60 | 60-76 | 60-76 |
| 6-9 years | 60-78 | 60-78 | 55-70 | 60-78 | 60-78 | 60-78 | 65-70 | 60-78 | 60-78 |
| 9-12 years | 70-82 | 60-82 | 55-70 | 70-82 | 70-82 | 70-82 | 70-75 | 70-82 | 70-82 |
| 12-18 years | 70-86 | 60-86 | 55-70 | 70-86 | 70-86 | 70-86 | 70-80 | 70-86 | 70-86 |

| | Temperature (C) | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Site<br>Age | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| Axillary | 36,1- | 35,9- | 36,3- | 36,3- | 36,3- | 36,3- | 36,3- | 36,3- | 36,3- |
| | 36,9 | 36,9 | 36,9 | 36,9 | 37,0 | 36,9 | 36,9 | 36,9 | 36,9 |
| Oral | 36,8- | 36,2- | 36,8- | 36,8- | 36,8- | 36,8- | 36,8- | 36,8- | 36,8- |
| | 37,3 | 37,3 | 37,3 | 37,3 | 37,3 | 37,3 | 37,3 | 37,3 | 37,3 |
| Rectal | 37,1- | 36,9- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- |
| | 37,9 | 37,9 | 37,7 | 37,7 | 38,0 | 37,7 | 37,7 | 37,7 | 37,7 |
| Tympanic | 36,1- | 36,5- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- | 37,3- |
| membrane | 36,9 | 37,5 | 37,7 | 37,7 | 37,7 | 37,7 | 37,7 | 37,7 | 37,7 |
| Skin /<br>Temporary<br>artery | 36,1-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 | 36,3-<br>36,9 |

Physical Examination will be summarized by subgroup (toilet trained, not toilet trained and overall).

# 4.4 Interim Analysis

No interim analysis is planned.

# 4.5 Data Safety Monitoring Board

Not applicable.

# 4.6 Safety Management Team

Not applicable.

# 5. DESCRIPTION OF NON-STANDARD DATA COLLECTED AND DERIVED VARIABLES

#### 5.1 Other Non-Standard Baseline Characteristics

Other baseline characteristic collected in the study is Main Diagnosis. The main Main Diagnosis data will be tabulated using descriptive statistics and listed.

#### 5.2 Non-Standard Disease History

Not applicable.

#### 5.3 Efficacy data

The efficacy data collected are:

- Information about diarrheal/watery stool/stool from Subjects Diary (domain SS);
- Global physician assessment at the end of treatment (domain QS).

#### 5.4 Non-standard Safety Data

The following non-standard safety data are collected: *Physical Examination (PE domain)*.

#### 5.5 Drug Accountability and Exposure

#### 5.5.1 Drug Accountability

Treatment compliance/drug accountability is defined as the number of sachets /capsules that were actually taken relative to the number of sachets /capsules that should have been taken for the duration of actual treatment exposure. The overall compliance, assessed by sachet/capsule count, will be calculated as follows:

#### 1. Racecadotril treatment:

 $\label{eq:compliance} \mbox{Compliance (\%)} = \frac{\mbox{Amount of ORS intake } * 100\%}{\mbox{[(Difference between Date/time of last dose and first dose in hours)/24 * Amount prescribed per day]}$ 

For prescribed ORS dose if frequency coded as "7=prn" (when necessary) then compliance will be stated as 100%, else the formula for compliance will be used.

The calculated percentage compliance will be categorized as:

- Too Low: < 80% compliance.
- Adequate:  $\geq 80\%$  to  $\leq 120\%$  compliance.
- Too High: > 120% compliance.

### 5.5.2 Exposure

Exposure analysis will be provided using EC domain. Descriptive statistics tables will be presented for:

- Mean duration of treatment<sup>1</sup> (in hours) by weight subgroups (less than 9 kg, from 9 kg to < 13 kg, from 13 kg to 27 kg, from more than 27 kg to 60 kg, 60 kg or higher) and overall;
- Mean duration of treatment (in hours) by age subgroup and overall;
- Cumulative dose divided by weight (mg/kg).

1 The duration of treatment will be assumed as 1 hour in case of single dose administration.

# 6. FURTHER SPECIFICATIONS TO THE STANDARD ANALYSES IN MODULE 2

#### 6.1 Trial Design [2]

#### **6.1.1** Trial Periods

The combination of trial arms and trial periods for the current trial is presented in the following diagram:

| | | Screening Period | Treatment Period | Follow-up Periods |
|---|---|---|---|---|
| Trial Arm A (RACE+ORS) | Subgroup<br>A | Screen | Racecadotril + ORS | Follow-up |
| | Subgroup<br>B | Screen | Racecadotril + ORS | Follow-up |
| | Subgroup<br>C | Screen | Racecadotril + ORS | Follow-up |
| Trial Arm B (ORS) | Subgroup<br>A | Screen | ORS | Follow-up |
| | Subgroup<br>B | Screen | ORS | Follow-up |
| | Subgroup<br>C | Screen | ORS | Follow-up |

Subgroups are defined by age categories:

- Subgroup A (from 3 to < 24 month)
- Subgroup B (from  $\geq$  2 to  $\leq$  12 years)
- Subgroup C (12 to < 18 years),

#### **6.1.2** Trial Elements

The start time of each intervention will be expressed relative to the first administration of investigational study drug closest to that intervention.

The Trial Elements are presented in the following diagram:

| Trial Element | Description of Element | <u> </u> | | Planned<br>Duration<br>of Element |
|---|---|---|---|---|
| Screen | Screening period | Date of<br>Informed<br>Consent | First dose of study treatment | |
| Racecadotril + ORS | Treatment period | First dose of<br>Racecadotril<br>+ ORS | Last dose of<br>Racecadotril + ORS | 5 days or less |
| ORS | Treatment period | First dose of ORS | Last dose of ORS | 5 days or<br>less |
| Follow-up | Safety<br>Follow-Up<br>period | Last dose of study treatment | Investigator's phone call 5-7 days after end of treatment visit | 5-7 days |

#### 6.1.3 Trial Arms

The trial arms for this study are made up of the following trial elements:

| | Elements | | | |
|---|---|---|---|---|
| Trial Arm | Screen | Racecadotril +<br>ORS | ORS | Follow-up |
| A | Y | Y | N | Y |
| В | Y | N | Y | Y |

#### 6.1.4 Visits and related definitions

Tests and examinations that were scheduled in the protocol will be related to the general time axis of the trial by relating the visit date on which a test or examination is performed to the start date of the trial element that describes the first administration of investigational study drug closest in time to the visit date of that test or examination (Reference Start Date/ Time).

| Test / Examination | Visit<br>name | Visit Label | Visit<br>Number | Reference<br>Start<br>Date/Time | Relative<br>Day<br>Number |
|---|---|---|---|---|---|
| Informed consent/assent | Screening | Screening | 1 | | |
| Randomization | Screening | Screening | 1 | | |
| Demographic data | Screening | Screening | 1 | | |

| Test / Examination | Visit<br>name | Visit Label | Visit<br>Number | Reference<br>Start<br>Date/Time | Relative<br>Day<br>Number |
|---|---|---|---|---|---|
| Medical history | Screening | Screening | 1 | | |
| Physical examination | Screening | Screening | 1 | | |
| In-or outpatient | Screening | Screening | 1 | | |
| Stool frequency within the last 24 hours | Screening | Screening | 1 | | |
| Inclusion/exclusion criteria | Screening | Screening | 1 | | |
| Vitals signs | Screening | Screening | 1 | | |
| Dispense study drug | Screening | Screening | 1 | | |
| Concomitant medication | Screening | Screening | 1 | | |
| Adverse events | Screening | Screening | 1 | | |
| Dispense diary | Screening | Screening | 1 | | |
| Collect diary | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |
| Physical examination | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |
| Compliance check | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |
| Adverse events | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |
| Collect study drug | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |

| Test / Examination | Visit<br>name | Visit Label | Visit<br>Number | Reference<br>Start<br>Date/Time | Relative<br>Day<br>Number |
|---|---|---|---|---|---|
| Concomitant medication | End of<br>Treatment | End of<br>Treatment | 2 | Date of last<br>dose of<br>study<br>treatment | Day 6 (*) |
| Adverse events | Follow-<br>Up | Safety follow-<br>up (phone call<br>5-7 days after<br>Visit 2) | 3 | Investigator 's phone call 5-7 days after end of treatment visit | Day 11-13 |
| Concomitant medication | Follow-<br>Up | Safety follow-<br>up (phone call<br>5-7 days after<br>Visit 2) | 3 | Investigator 's phone call 5-7 days after end of treatment visit | Day 11-13 |

<sup>(\*)</sup> or within 24 h after recovery if this occurs before day 6

# 6.2 Further Specifications to the Standard Tables in Module 2

Not applicable.

# 6.3 Other Further Specifications

Not applicable.

# 7. CHANGES TO PLANNED ANALYSES

No changes will be made to the final SAP

# 8. REFERENCE

- 1. Abbott SAP Module 2
- 2. CDISC terminology, see <a href="http://www.cdisc.org">http://www.cdisc.org</a>.

#### 9. APPENDICES

#### 9.1 Study Flowchart

Note: Any additional medical procedures not included into this study protocol can be performed within routine clinical practice in each medical institution.

| Period | Screening | End of Treatment period | Safety follow-up<br>(phone call 5-7 days<br>after Visit 2) |
|---|---|---|---|
| Visit | 1 | 2 | 3 |
| Day | 1 | 6 <sup>2</sup> | 11-13 |
| Informed consent | X | | |
| Randomization | X | | |
| Demographic data | X | | |
| Medical history | X | | |
| Pregnancy Test <sup>4</sup> | X | | |
| Physical examination <sup>3</sup> | X | X | |
| In- or outpatient | X | | |
| Stool frequency within the last 24 hours | X | | |
| Inclusion/exclusion criteria | X | | |
| Vitals signs | X | X | |
| Dispense study drug | X | | |
| Concomitant medication | X | X | X if applicable |
| Compliance check | | X | |
| Adverse events | X | X | X |
| Collect study drug | | X | |
| Dispense diary | $X^{1}$ | | |
| Collect diary | | X | |

<sup>&</sup>lt;sup>1</sup> Subjects' parent/caregivers have to fill in their daily diaries continuously.

<sup>&</sup>lt;sup>2</sup> or within 24 h after recovery if this occurs before day 6

<sup>&</sup>lt;sup>3</sup> including assessment of dehydration level

<sup>&</sup>lt;sup>4</sup> for females of child-bearing potential, urine test

# 9.2 Tables, Listings and Figures

#### **9.2.1** Tables

For the shells of the non-standard tables, see Section 10.1.

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| DST001 | Subject Disposition | 10.1.1.1 | Subject Disposition - All<br>Subjects Allocated to<br>Treatment Subject Sample | | | |
| DVT001 | Protocol Deviations | 10.1.1.2 | Protocol Deviations – All<br>Subjects Allocated to<br>Treatment Subject Sample | | | |
| DVT002 | Protocol Deviations | 10.1.1.3 | Subject Samples - All<br>Subjects Allocated to<br>Treatment Subject Sample | | | |
| DMT002 | Demographic Data | 10.1.1.5 | Demographics – Safety<br>Sample | | | |
| DMT002 | Demographic Data | 10.1.1.6 | Demographics –Full Analysis<br>Subject Sample | | | |
| VST003 | Vital Signs | 10.1.1.8 | Other Baseline Characteristics – Safety Sample | | | |
| VST003 | Vital Signs | 10.1.1.9 | Other Baseline Characteristics – Full Analysis Subject Sample | | | |
| MHT001 | Medical History | 10.1.1.10 | Medical History – All<br>Subjects Allocated to<br>Treatment Subject Sample | | | |
| MHT001 | Medical History | 10.1.1.11 | Medical History – Safety<br>Sample | | | |
| MHT001 | Medical History | 10.1.1.12 | Medical History – Full<br>Analysis Subject Sample | | | |
| NST001 | Medical History | 10.1.1.13 | Main Diagnosis - All Subjects<br>Allocated to Treatment<br>Subject Sample | | | |
| NST002 | Medical History | 10.1.1.14 | Main Diagnosis - Safety<br>Sample | | | |
| NST003 | Medical History | 10.1.1.15 | Main Diagnosis - Full<br>Analysis Subject Sample | | | |
| CMT001 | Concomitant<br>Medications | 10.1.1.16 | Concomitant Medications –<br>All Subjects Allocated to<br>Treatment Subject Sample | | | |
| CMT001 | Concomitant<br>Medications | 10.1.1.17 | Concomitant Medications –<br>Safety Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| CMT001 | Concomitant<br>Medications | 10.1.1.18 | Concomitant Medications –<br>Full Analysis Subject Sample | | | |
| DAT001 | Treatment<br>Compliance | 10.1.1.19 | Compliance to Study Drug –<br>All Subjects Allocated to<br>Treatment Subject Sample | | | |
| DAT001 | Treatment<br>Compliance | 10.1.1.20 | Compliance to Study Drug –<br>Safety Sample | | | |
| DAT001 | Treatment<br>Compliance | 10.1.1.21 | Compliance to Study Drug –<br>Full Analysis Subject Sample | | | |
| AET001 | Adverse Events | 10.1.3.1.1 | Overall Summary of Adverse<br>Events – Safety Sample | | | |
| AET002 | Adverse Events | 10.1.3.1.2 | Incidence of TEAEs – Safety<br>Sample | | | |
| AET005 | Adverse Events | 10.1.3.1.3 | Incidence of TEAEs With a<br>Reasonable Possibility for a<br>Causal Relationship<br>(Investigator's Judgment) –<br>Safety Sample | | | |
| AET006 | Adverse Events | 10.1.3.1.4 | Incidence of TEAEs by Maximum Severity (Investigator's Judgment) – Safety Sample | | | |
| AET007 | Adverse Events | 10.1.3.1.5 | Incidence of TESAEs –<br>Safety Sample | | | |
| AET008 | Adverse Events | 10.1.3.1.6 | Incidence of TEAEs Leading<br>to Study Termination – Safety<br>Sample | | | |
| VST001 | Vital Signs | 10.1.3.2.1 | Summary of Vital Signs –<br>Safety Sample | | | |
| VST002 | Vital Signs | 10.1.3.2.2 | Incidence of Markedly<br>Abnormal Vital Signs –<br>Safety Sample | | | |
| NST004 | Physical<br>Examination | 10.1.3.3.1 | Physical Examination by subgroup (Toilet trained / Not toilet trained) – Safety Sample | | | |
| NST005 | Exposure | 10.1.3.4.1 | Treatment duration – Safety<br>Sample | | | |
| NST006 | Exposure | 10.1.3.4.2 | Cumulative dose by weight (mg/kg) – Safety Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST007 | Subject Status | 10.1.4.1.1 | Duration of diarrhea: time to<br>last diarrheal/watery stool<br>before recovery by days.<br>Kaplan-Meier analysis – Full<br>Analysis Subject Sample | | | |
| NST008 | Subject Status | 10.1.4.1.2.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample | | | |
| NST009 | Subject Status | 10.1.4.1.2.2 | Duration of diarrhea. Cox<br>Regression Model – Full<br>Analysis Subject Sample | | | |
| NST010 | Subject Status | 10.1.4.1.3.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Full Analysis Subject Sample | | | |
| NST011 | Subject Status | 10.1.4.1.3.2 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Full Analysis Subject Sample | | | |
| NST012 | Subject Status | 10.1.4.1.3.3 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Full Analysis Subject Sample | | | |
| NST013 | Subject Status | 10.1.4.1.3.4 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants less than 9 kg – Full Analysis Subject Sample | | | |
| NST014 | Subject Status | 10.1.4.1.3.5 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants from 9 kg to < 13 kg – Full Analysis Subject Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST015 | Subject Status | 10.1.4.1.3.6 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from 13 kg to 27 kg – Full Analysis Subject Sample | | | |
| NST016 | Subject Status | 10.1.4.1.3.7 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from more than 27 kg to 60 kg – Full Analysis Subject Sample | | | |
| NST017 | Subject Status | 10.1.4.1.3.8 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children or adolescents of 60 kg or higher – Full Analysis Subject Sample | | | |
| NST018 | Subject Status | 10.1.4.1.3.9 | Duration of diarrhea. Number<br>of stools during the study -<br>Full Analysis Subject Sample | | | |
| NST019 | Subject Status | 10.1.4.1.4 | Duration of diarrhea: time to<br>last diarrheal/watery stool<br>before recovery by days.<br>Kaplan-Meier analysis – Per<br>Protocol Subject Sample | | | |
| NST020 | Subject Status | 10.1.4.1.5.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results – Per Protocol Subject Sample | | | |
| NST021 | Subject Status | 10.1.4.1.5.2 | Duration of diarrhea. Cox<br>Regression Model – Per<br>Protocol Subject Sample | | | |
| NST022 | Subject Status | 10.1.4.1.6.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Per Protocol Subject Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST023 | Subject Status | 10.1.4.1.6.2 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Per Protocol Subject Sample | | | |
| NST024 | Subject Status | 10.1.4.1.6.3 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Per Protocol Subject Sample | | | |
| NST025 | Subject Status | 10.1.4.1.6.4 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants less than 9 kg – Per Protocol Subject Sample | | | |
| NST026 | Subject Status | 10.1.4.1.6.5 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants from 9 kg to < 13 kg – Per Protocol Subject Sample | | | |
| NST027 | Subject Status | 10.1.4.1.6.6 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from 13 kg to 27 kg – Per Protocol Subject Sample | | | |
| NST028 | Subject Status | 10.1.4.1.6.7 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from more than 27 kg to 60 kg – Per Protocol Subject Sample | | | |
| NST029 | Subject Status | 10.1.4.1.6.8 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children or adolescents of 60 kg or higher – Per Protocol Subject Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST030 | Subject Status | 10.1.4.1.6.9 | Duration of diarrhea. Number<br>of stools during the study -<br>Per Protocol Subject Sample | | | |
| NST031 | Subject Status | 10.1.4.1.7 | Number of stools per day<br>(toilet trained subgroup) –<br>Full Analysis Subject Sample | | | |
| NST032 | Subject Status | 10.1.4.1.8 | Number of watery stools per<br>day (toilet trained subgroup) –<br>Full Analysis Subject Sample | | | |
| NST033 | Subject Status | 10.1.4.1.9 | Cumulative number of stools<br>until recovery or end of<br>treatment by days – Full<br>Analysis Subject Sample | | | |
| NST034 | Subject Status | 10.1.4.2.1 | Time to recovery: time to evacuation of the first of two consecutive normal stools or no stool after first normal stool within 12 hours by days. Kaplan-Meier analysis – Full Analysis Subject Sample | | | |
| NST035 | Subject Status | 10.1.4.2.2.1 | Time to recovery. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample | | | |
| NST036 | Subject Status | 10.1.4.2.2.2 | Time to recovery. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample | | | |
| NST037 | Subject Status | 10.1.4.2.2.3 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Full Analysis Subject Sample | | | |
| NST038 | Subject Status | 10.1.4.2.2.4 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Full Analysis Subject Sample | | | |
| NST039 | Subject Status | 10.1.4.2.2.5 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Full Analysis Subject Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST040 | Subject Status | 10.1.4.2.2.6 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Infants less than 9 kg – Full Analysis Subject Sample | | | |
| NST041 | Subject Status | 10.1.4.2.2.7 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Infants from 9 kg to < 13 kg – Full Analysis Subject Sample | | | |
| NST042 | Subject Status | 10.1.4.2.2.8 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children from 13 kg to 27 kg – Full Analysis Subject Sample | | | |
| NST043 | Subject Status | 10.1.4.2.2.9 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children from more than 27 kg to 60 kg – Full Analysis Subject Sample | | | |
| NST044 | Subject Status | 10.1.4.2.2.10 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children or adolescents of 60 kg or higher – Full Analysis Subject Sample | | | |
| NST045 | Questionnaires | 10.1.4.2.3 | Global Physician Assessment<br>at the end of treatment – Full<br>Analysis Subject Sample | | | |
| NST046 | Questionnaires | 10.1.4.2.4.1 | Global Physician Assessment<br>at the end of treatment for<br>weight/dosing category<br>Infants less than 9 kg – Full<br>Analysis Subject Sample | | | |

| | | | | Produced for | | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| NST047 | Questionnaires | 10.1.4.2.4.2 | Global Physician Assessment<br>at the end of treatment for<br>weight/dosing category<br>Infants from 9 kg to < 13 kg –<br>Full Analysis Subject Sample | | | |
| NST048 | Questionnaires | 10.1.4.2.4.3 | Global Physician Assessment<br>at the end of treatment for<br>weight/dosing category<br>Children from 13 kg to 27 kg<br>– Full Analysis Subject<br>Sample | | | |
| NST049 | Questionnaires | 10.1.4.2.4.4 | Global Physician Assessment<br>at the end of treatment for<br>weight/dosing category<br>Children from more than 27<br>kg to 60 kg – Full Analysis<br>Subject Sample | | | |
| NST050 | Questionnaires | 10.1.4.2.4.5 | Global Physician Assessment<br>at the end of treatment for<br>weight/dosing category<br>Children or adolescents of 60<br>kg or higher – Full Analysis<br>Subject Sample | | | |

# 9.2.2 Listings

For the shells of the non-standard listings, see Section 10.2.

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| DSL001 | Subject Disposition | 12.2.1.1 | Subjects Who Prematurely Terminated the Study Prior to Treatment Allocation - All Subjects Consented Subject Sample | | | |
| DSL002 | Subject Disposition | 12.2.1.2 | Subjects Allocated to Treatment - All Subjects Allocated to Treatment Subject Sample | | | |
| DSL003 | Subject Disposition | 12.2.1.3 | Subjects Allocated to Treatment<br>Who Prematurely Terminated<br>the Study - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |

| | | | | Produced | for: | |
|---|---|---|---|---|---|---|
| Output<br>Code | Clinical Domain | Output<br>Number | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| DVL001 | Protocol Deviations | 12.2.2.1 | Subjects With Protocol<br>Deviations - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |
| IEL002 | Inclusion/Exclusion | 12.2.2.2 | Subjects With Deviations from<br>Inclusion or Exclusion Criteria -<br>All Subjects Consented Subject<br>Sample | | | |
| DVL002 | Protocol Deviations | 12.2.3.1 | Subjects Excluded From the<br>Subject Samples - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |
| DML002 | Demographic Data | 12.2.4.1 | Demographics - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |
| NSL001 | Vital Signs | 12.2.4.2 | Other Baseline Characteristics -<br>All Subjects Allocated to<br>Treatment Subject Sample | | | |
| NSL002 | Reproductive<br>System Findings | 12.2.4.3 | Urinary Pregnancy Test / Childbearing Potential - All Subjects Allocated to Treatment Subject Sample | | | |
| MHL001 | Medical History | 12.2.4.4 | Medical History: General - All<br>Subjects Allocated to Treatment<br>Subject Sample | | | |
| MHL002 | Medical History | 12.2.4.5 | Medical History: MedDRA<br>Coding - All Subjects Allocated<br>to Treatment Subject Sample | | | |
| CML001 | Concomitant<br>Medications | 12.2.4.6 | Concomitant Medication:<br>General - All Subjects Allocated<br>to Treatment Subject Sample | | | |
| CML002 | Concomitant<br>Medications | 12.2.4.7 | Concomitant Medication: WHO-<br>DD Coding - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |
| NSL003 | Medical History | 12.2.4.7 | Main Diagnosis - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |
| DAL001 | Drug Accountability | 12.2.5.1 | Drug Accountability and<br>Compliance - All Subjects<br>Allocated to Treatment Subject<br>Sample | | | |

| Output<br>Code | Clinical Domain | Output<br>Number | | Produced | for: | for: |
|---|---|---|---|---|---|---|
| | | | Title | Headline<br>Results | SMT | Interim<br>Analysis |
| AEL008 | Adverse Events | 12.2.7.1 | AEs: General - All Subjects<br>Consented Subject Sample | | | |
| AEL002 | Adverse Events | 12.2.7.2 | AEs: MedDRA Coding - All<br>Subjects Consented Subject<br>Sample | | | |
| AEL010 | Adverse Events | 10.1.3.1.9 | Listing of Other SAEs - All<br>Subjects Consented Subject<br>Sample | | | |
| AEL011 | Adverse Events | 10.1.3.1.11 | Listing of TEAEs Leading to<br>Study Termination – Safety<br>Sample | | | |
| AEL012 | Adverse Events | 10.1.3.1.12 | Listing of TEAEs Leading to Discontinuation of Study Drug – Safety Sample | | | |
| VSL004 | Vital Signs | 12.2.8.8 | Markedly Abnormal Vital Signs – Safety Sample | | | |
| VSL005 | Vital Signs | 12.2.8.9 | Vital Signs - All Subject<br>Allocated to Treatment Subject<br>Sample | | | |
| SVL001 | Subject Visits | 12.2.8.15 | Subject Visits – All Subject<br>Allocated to Treatment Subject<br>Sample | | | |
| NSL004 | Physical<br>Examination | 12.2.9.1 | Physical Examination - All<br>Subject Allocated to Treatment<br>Subject Sample | | | |
| NSL005 | Questionnaries | 12.2.9.2 | Global Physician Assessment -<br>All Subject Allocated to<br>Treatment Subject Sample | | | |
| NSL006 | Subject Status | 12.2.9.3 | Stool Evacuation- All Subject<br>Allocated to Treatment Subject<br>Sample | | | |

# 9.2.3 Figures

For the shells of the non-standard figures, see Section 10.3.

| Output<br>Code | Clinical Domain | Output<br>Number | | Produced for: | | |
|---|---|---|---|---|---|---|
| | | | Title | Headline results | SMT | Interim<br>analysis |
| DSF001 | Subject Disposition | 10.1.4.1 | Flowchart of Subject Disposition | | | |
| DSF002 | Subject Disposition | 10.1.4.2 | Flowchart of Subject samples | | | |
| NSF001 | Subject Status | 10.1.4.1.1 | Kaplan-Meier Plot of duration of<br>diarrhea – Full Analysis Subject<br>Sample | | | |
| NSF002 | Subject Status | 10.1.4.1.2 | Kaplan-Meier Plot of duration of<br>diarrhea— Per Protocol Subject<br>Sample | | | |
| NSF003 | Subject Status | 10.1.4.1.3 | Kaplan-Meier Plot for time to<br>recovery – Full Analysis Subject<br>Sample | | | |

# 9.3 Non-standard Tables, Listings and Figures Shells

# 9.3.1 Non-Standard Tables

| Table code | Comment |
|---|---|
| 10.1.1.13 | Main Diagnosis – All Subjects Allocated to Treatment Subject Sample |
| 10.1.1.14 | Main Diagnosis – Safety Sample |
| 10.1.1.15 | Main Diagnosis – Full Analysis Subject Sample |
| 10.1.3.3.1 | Physical Examination by subgroup (Toilet trained / Not toilet trained) – Safety Sample |
| 10.1.3.4.1 | Treatment duration – Safety Sample |
| 10.1.3.4.2 | Cumulative dose by weight (mg/kg) – Safety Sample |
| 10.1.4.1.1 | Duration of diarrhea: time to last diarrheal/watery stool before recovery by days. Kaplan-Meier analysis – Full Analysis Subject Sample |
| 10.1.4.1.2.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample |
| 10.1.4.1.2.2 | Duration of diarrhea. Cox Regression Model – Full Analysis Subject Sample |
| 10.1.4.1.3.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Full Analysis Subject Sample |
| 10.1.4.1.3.2 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Full Analysis Subject Sample |
| 10.1.4.1.3.3 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Full Analysis Subject Sample |
| 10.1.4.1.3.4 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants less than 9 kg – Full Analysis Subject Sample |
| 10.1.4.1.3.5 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants from 9 kg to < 13 kg - Full Analysis Subject Sample |
| 10.1.4.1.3.6 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from 13 kg to 27 kg – Full Analysis Subject Sample |

10.1.4.1.6.9

Protocol no. RACE3003

06 Aug 18

| , | $\sim$ |
|---|---|
| 10.1.4.1.3.7 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from more than 27 kg to 60 kg – Full Analysis Subject Sample |
| 10.1.4.1.3.8 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children or adolescents of 60 kg or higher – Full Analysis Subject Sample |
| 10.1.4.1.3.9 | Duration of diarrhea. Number of stools during the study - Full Analysis Subject Sample |
| 10.1.4.1.4 | Duration of diarrhea: time to last diarrheal/watery stool before recovery by days. Kaplan-Meier analysis – Per Protocol Subject Sample |
| 10.1.4.1.5.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results – Per Protocol Subject Sample |
| 10.1.4.1.5.2 | Duration of diarrhea. Cox Regression Model – Per Protocol Subject Sample |
| 10.1.4.1.6.1 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Per Protocol Subject Sample |
| 10.1.4.1.6.2 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Per Protocol Subject Sample |
| 10.1.4.1.6.3 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Per Protocol Subject Sample |
| 10.1.4.1.6.4 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants less than 9 kg – Per Protocol Subject Sample |
| 10.1.4.1.6.5 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category infants from 9 kg to < 13 kg – Per Protocol Subject Sample |
| 10.1.4.1.6.6 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from 13 kg to 27 kg – Per Protocol Subject Sample |
| 10.1.4.1.6.7 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children from more than 27 kg to 60 kg – Per Protocol Subject Sample |
| 10.1.4.1.6.8 | Duration of diarrhea. Descriptive statistics (in hours) and comparison results for weight/dosing category children or adolescents of 60 kg or higher – Per Protocol Subject Sample |

Duration of diarrhea. Number of stools during the study - Per Protocol Subject Sample

Protocol no. RACE3003

06 Aug 18

| 10.1.4.1.7 | Number of stools per day (toilet trained subgroup) – Full Analysis Subject Sample |
|---|---|
| 10.1.4.1.8 | Number of watery stools per day (toilet trained subgroup) – Full Analysis Subject Sample |
| 10.1.4.1.9 | Cumulative number of stools until recovery or end of treatment by days – Full Analysis Subject Sample |
| 10.1.4.2.1 | Time to recovery: time to evacuation of the first of two consecutive normal stools or no stool after first normal stool within 12 hours by days. Kaplan-Meier analysis – Full Analysis Subject Sample |
| 10.1.4.2.2.1 | Time to recovery. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample |
| 10.1.4.2.2.2 | Time to recovery. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample |
| 10.1.4.2.2.3 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from 3 to < 24 month – Full Analysis Subject Sample |
| 10.1.4.2.2.4 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from >= 2 to <12 years – Full Analysis Subject Sample |
| 10.1.4.2.2.5 | Time to recovery. Descriptive statistics (in hours) and comparison results for age group from 12 to < 18 years – Full Analysis Subject Sample |
| 10.1.4.2.2.6 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Infants less than 9 kg – Full Analysis Subject Sample |
| 10.1.4.2.2.7 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Infants from 9 kg to < 13 kg – Full Analysis Subject Sample |
| 10.1.4.2.2.8 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children from 13 kg to 27 kg – Full Analysis Subject Sample |
| 10.1.4.2.2.9 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children from more than 27 kg to 60 kg – Full Analysis Subject Sample |
| 10.1.4.2.2.10 | Time to recovery. Descriptive statistics (in hours) and comparison results for weight/dosing category Children or adolescents of 60 kg or higher – Full Analysis Subject Sample |
| 10.1.4.2.1 | Time to recovery: time to evacuation of the first of two consecutive normal stools or no stool after first normal stool within 12 hours by days. Kaplan-Meier analysis – Full Analysis Subject Sample |
| 10.1.4.2.2 | Time to recovery. Descriptive statistics (in hours) and comparison results – Full Analysis Subject Sample |

Protocol no. RACE3003

06 Aug 18

| 10.1.4.2.3 | Global Physician Assessment at the end of treatment – Full Analysis Subject Sample |
|---|---|
| 10.1.4.2.4.1 | Global Physician Assessment at the end of treatment for weight/dosing category Infants less than 9 kg – Full Analysis Subject Sample |
| 10.1.4.2.4.2 | Global Physician Assessment at the end of treatment for weight/dosing category Infants from 9 kg to < 13 kg – Full Analysis Subject Sample |
| 10.1.4.2.4.3 | Global Physician Assessment at the end of treatment for weight/dosing category Children from 13 kg to 27 kg – Full Analysis Subject Sample |
| 10.1.4.2.4.4 | Global Physician Assessment at the end of treatment for weight/dosing category Children from more than 27 kg to 60 kg – Full Analysis Subject Sample |
| 10.1.4.2.4.5 | Global Physician Assessment at the end of treatment for weight/dosing category Children or adolescents of 60 kg or higher – Full Analysis Subject Sample |